CLINICAL TRIAL: NCT05621044
Title: Smartphone App to Increase and Maintain Physical Activity in African American Men (FitBrothers) Phase II
Brief Title: Physical Activity Smartphone App for African American Men (FitBros) Ph II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: Pennington Biomedical Research Center (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0340; 4R42MD014947-02 (NIH)
Record Dates: First submitted 2022-11-10; First posted 2022-11-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Exercise; Health Behavior; Technology
MeSH Terms: conditions — Motor Activity; Health Behavior

STUDY DESIGN:
Intervention Model Description: Behavioral
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FitBrothers smartphone active app (Experimental): Participants will be expected to engage with the FitBrothers app on a daily basis. Daily alerts and notifications will engage users in daily use of the app and provide up-to-date information on users' progress. Participant responses will also be used to evaluate additional or on-going support of users' needs (e.g., increase/ decrease prompts based on user preferences, tailored messages around a set goal, etc.). To protect privacy and to ensure that the participant is the person completing the app activities, KB will uniquely identify the user's smartphone based off the device's "hardware footprint". The app will upload all app activity data to the KB secured web server database.
  Interventions: Behavioral: FitBrothers smartphone active app
- Comparator app (Active Comparator): Nike Training Club is a free app available on iOS and Android platforms. The app is designed to increase fitness in users through a variety of mechanisms. Similar to FitBrothers, men will be able to track and monitor their physical activity level, set goals, engage in competitions, and upload activity data from a wearable. They will also be provided with preset workouts, receive guidance from an expert, and receive personalized plans that automatically adapt to user behavior. Unlike the FitBrothers app, the Nike Training Club app was not developed with input from African American men, does not track health information (e.g. blood pressure, blood glucose), does not have a theoretical basis, and does not have specific strategies for maintenance.
  Interventions: Behavioral: Nike Training Club

INTERVENTIONS:
Behavioral: FitBrothers smartphone active app — The FitBrothers smartphone active app is designed to assist African American men with adopting and maintaining PA. The app will be developed with significant input from African American men and contain self-monitoring, goal setting, reward, and educational components. The app will include additional elements including PA adoption strategies, competitions, incentives, health information, and greater compatibility with activity monitoring devices. The intervention is based on the Social Cognitive and Self-Determination theories and is culturally tailored.
  Arms: FitBrothers smartphone active app
Behavioral: Nike Training Club — The app is designed to increase fitness in users through a variety of mechanisms. Users are able to track and monitor their physical activity level, set goals, engage in competitions, and upload activity data from a wearable. They will also be provided with preset workouts, receive guidance from an expert, and receive personalized plans that automatically adapt to user behavior.
  Arms: Comparator app

SUMMARY:
Low physical activity levels contribute to African American men experiencing health disparities across a number of chronic diseases. Studies have been effective in increasing physical activity levels in African American men; but few have targeted maintenance of behavior change and none have utilized emerging technologies. The purpose of the current study is to further develop a mobile phone application for African American men that will help them initiate and maintain their physical activity levels.

DETAILED DESCRIPTION:
Physical activity (PA) is a modifiable risk factor for a number of preventable chronic diseases, including cardiovascular disease, strokes, obesity, and diabetes. These conditions constitute health disparities for African American men. Behavioral interventions have proven to be effective in promoting increases in physical activity. While behavior change programs have been shown to assist participants in sustaining behavior change, very few programs have specifically targeted African American men. The use of mHealth, as opposed to other avenues of intervention delivery, is based on published reports documenting that African Americans perceive mobile technology as an acceptable means of intervention delivery. In addition, ownership of smartphones and the use of text messaging are highest among African Americans compared to other ethnic groups. Therefore, a mHealth intervention targeting African American men seems feasible and potentially effective. Our preliminary data show that a PA maintenance smartphone app for African American men that contains self-monitoring, goal-setting, reinforcement, and behavioral lessons was well received by this population. However, the qualitative data revealed that the men believed additional components were necessary to fully tailor the app for African American men, including personalization, chronic disease health information, dietary information, competition, and incentives. In addition, the investigators will tailor the intervention to the sociocultural needs of African American men. The purpose of the Fast-Track STTR is to incorporate these elements within an existing smartphone app. The FitBrothers app was developed through a Phase I consisting of (1) iterative focus groups, (2) developing a conceptual model, and (3) conducting beta testing and this Phase II will consist of (1) developing a full-scale FitBrothers app, (2), conducting usability testing, and (3) conducting a comparative effectiveness trial to assess the effectiveness of the app compared to a similar, well-known app in the marketplace. To our knowledge, no study has utilized mobile phones as a means of effecting PA levels in African American men. FitBrothers will address an unmet need in the marketplace as it will be the first smartphone app that is targeted toward PA adoption and maintenance in African American men. The fact that mHealth is acceptable to- and the fact that the application will be developed in collaboration with African American men, leads us to hypothesize that African American men will view the mHealth intervention as acceptable, feasible, and effective. The Fast-Track STTR project will be led by a team that has worked together previously and includes researchers and multimedia developers from Klein Buendel, Inc. (KB), Georgetown University, and Pennington Biomedical Research Center.

ELIGIBILITY:
Comparative Effectiveness Trial (CET) Inclusion criteria:

* self-identified African American male
* at least 30 years of age
* BMI > 18.5 kg/m2 and < 45 kg/m2
* resting systolic blood pressure # 159 mmHg and a diastolic blood pressure # 99 (to reduce risk of exercise-induced cardiovascular events)
* free of significant medical problems that would impact their ability to engage in aerobic and/or resistance training
* owns a smartphone
* sedentary at baseline (not being physically active ≥3 d·wk-1 for 20 min each time for the previous 6 months, not participating in regular resistance exercise, and having an average daily accelerometer step count less than the 50th percentile for age and gender).

Comparative Effectiveness Trial (CET) Exclusion criteria:

* unwilling to give written informed consent
* conditions that prevent regular exercise
* conditions that the medical or principal investigator determine to warrant exclusion

Min Age: 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-01-22 (Actual); Study Completion 2026-01-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Physical activity-Acti Graph at 9 Months | Baseline and 9 months
  Steps per day will be collected using the ActiGraph WGT3X+BT accelerometer. The device is worn on the wrist for a 7-day period.

SECONDARY OUTCOMES:
Change from Baseline in Weight at 9 Months | Baseline and 9 months
  Weight of each participant will be measured with a scale.
Change from Baseline in Blood Pressure at 9 months | Baseline and 9 months
  Systolic and diastolic blood pressure will be measured at rest, under highly-controlled conditions. All blood pressure measurements will be obtained using a Colin STBP-780 automated blood pressure monitor. The first value will be discarded and the average of the last 3 values will be used, per standard Pennington Biomedical Research Center (PBRC) procedures.
Change from Baseline in Quality of Life Assessment at 9 Months | Baseline and 9 months
  The SF-36 Short Form Health Survey (SF-36) questionnaire will assess quality of life in a number of physiological and mental health domains.
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Change from Baseline in Dietary Habits at 9 Months | Baseline and 9 months
  The National Cancer Institute's Automated Self-Administered 24-hour Recall will be used to estimate daily intake of selected nutrients and macronutrients, food group servings, and alcohol.
  The NCI's Automated Self-Administered 24-hour Recall (ASA24) will be used to estimate daily intake of nutrients and macronutrients, food group servings, and alcohol. This tool enables self-administered 24-hour dietary recalls and calculates Healthy Eating Index scores (minimum score=0, maximum score=100). Healthy Eating Index measures diet quality and assesses conformance to federal dietary guidance. Higher scores reflect better dietary habits.
Satisfaction Assessment | 9 months
  A questionnaire will be used to assess each participant's satisfaction with the FitBrothers app.
  The questionnaire will assess satisfaction, helpfulness, enjoyment, and relevance across all components of app. Mean scores of 3.5 or greater, rated on a scale of 1 (poor) to 5 (excellent), will be deemed acceptable.
System Usability Scale (SUS) | 9 months
  The System Usability Scale (SUS) is a validated, 10-item measure provides a global view of subjective usability for technology. The 10 questions have 5 response options from "strongly disagree" to "strongly agree". SUS yields a single number representing a composite measure of the overall usability of the system being studied. Note that scores for individual items are not meaningful on their own. To calculate the SUS score the score contributions from each item are summed. Each item's score contribution ranges from 0 to 4. For items 1,3,5,7,and 9 the score contribution is the scale position minus 1. For items 2,4,6,8 and 10, the contribution is 5 minus the scale position. The sum of these scores are multiplied by 2.5 to obtain the overall value of SU.SUS scores have a range of 0 to 100. SUS scores > 68 are considered acceptable.
FitBrothers App Usage | 9 months
  FitBrothers app usage will be assessed via a number of app usage sessions. Usage will be collected using Webtrends.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Newton, PHD, Principal Investigator — Pennington Biomedical Research Center
Locations (3):
- United States (3):
  - Klein Buendel, Inc., Golden, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana

REFERENCES:
- [Derived] Nuss K, Brice A, Hebert C, Nauta P, Stull AJ, Swift DL, Griffith DM, Buller DB, Newton RL Jr. A Culturally Tailored mHealth Intervention (MobileMen App) to Promote Physical Activity in African American Men: Protocol for a Comparative Effectiveness Trial. JMIR Res Protoc. 2025 Jul 4;14:e67809. doi: 10.2196/67809. PMID 40613599